CLINICAL TRIAL: NCT05867810
Title: Nutritional Status Among Upper Gastrointestinal Cancer Patients Upon Admission
Acronym: RSCH ID-22-012
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, ChiouYi Ho, Dietitian, Universiti Putra Malaysia
Other Study IDs: NMRR ID-22-00792-HKU; RSCH ID-22-01272-6KC (Other: Ministry of Health Medical Research and Ethics Committee (MREC))
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Upper Gastrointestinal Cancer Patients Upon Admission; Nutritional Status
Keywords: Upper Gastrointestinal Cancer Patients; upon admission; Nutritional Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross-sectional study. Data on clinical, anthropometric, biochemical profile and dietary intake Upper Gastrointestinal Cancer Patients upon admission are traced and collected.

DETAILED DESCRIPTION:
As per routine care, on the day of admission, nutrition assessment and clinical examination of all in-patients will be carried out. Patient screening will be done by assigned investigator based on the dietitian censes based on inclusion and exclusion criteria. The investigator will trace the data from medical system and record in the data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Admitted UGIC patient
* Seen by dietitian in ward

Exclusion Criteria:

* Not admitted in ward
* Aged <18 years old
* Non-Malaysian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: histologically confirmed Upper Gastrointestinal Cancers
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
nutrition assessment | within 2 hours upon admission
  anthropometry (weight)
nutrition assessment | within 24 hours upon admission
  dietary assessment
nutrition assessment | within 24 hours upon admission
  nutrition impact symptom (NIS)
nutrition assessment | within 24 hours upon admission
  subjective global assessment (SGA)

SECONDARY OUTCOMES:
Biochemical data | within 2 hours upon admission
  albumin
Biochemical data | within 2 hours upon admission
  lymphocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Kanser Negara (National Cancer Institute), Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Reber E, Schonenberger KA, Vasiloglou MF, Stanga Z. Nutritional Risk Screening in Cancer Patients: The First Step Toward Better Clinical Outcome. Front Nutr. 2021 Apr 7;8:603936. doi: 10.3389/fnut.2021.603936. eCollection 2021. PMID 33898493
- [Background] Ho CY, Ibrahim Z, Abu Zaid Z, Mat Daud Z', Md Yusop NB. Clinical malnutrition predictive model among gynecologic cancer patients prior to elective operation: A cross-sectional study. Clin Nutr. 2021 Jun;40(6):4373-4379. doi: 10.1016/j.clnu.2021.01.008. Epub 2021 Jan 12. PMID 33485706
- [Background] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Background] Chen MJ, Wu IC, Chen YJ, Wang TE, Chang YF, Yang CL, Huang WC, Chang WK, Sheu BS, Wu MS, Lin JT, Chu CH. Nutrition therapy in esophageal cancer-Consensus statement of the Gastroenterological Society of Taiwan. Dis Esophagus. 2018 Aug 1;31(8). doi: 10.1093/dote/doy016. PMID 29860406
- [Background] Allum W, Lordick F, Alsina M, Andritsch E, Ba-Ssalamah A, Beishon M, Braga M, Caballero C, Carneiro F, Cassinello F, Dekker JW, Delgado-Bolton R, Haustermans K, Henning G, Hutter B, Lovey J, Netikova IS, Obermannova R, Oberst S, Rostoft S, Saarto T, Seufferlein T, Sheth S, Wynter-Blyth V, Costa A, Naredi P. ECCO essential requirements for quality cancer care: Oesophageal and gastric cancer. Crit Rev Oncol Hematol. 2018 Feb;122:179-193. doi: 10.1016/j.critrevonc.2017.12.019. Epub 2018 Jan 2. PMID 29458786
- [Background] Deftereos I, Hitch D, Butzkueven S, Carter V, Arslan J, Fetterplace K, Fox K, Ottaway A, Pierce K, Steer B, Varghese J, Kiss N, Yeung J. Implementation of a standardised perioperative nutrition care pathway in upper gastrointestinal cancer surgery: A multisite pilot study. J Hum Nutr Diet. 2023 Apr;36(2):479-492. doi: 10.1111/jhn.13018. Epub 2022 May 18. PMID 35441757
- [Background] Azizah A, Hashimah B, Siti Zubaidah A, Puteri N, Nabihah A, Sukumaran R, et al. Malaysian National Cancer Registry Report (MNCR) 2012-2016. 2019.
- [Background] Deftereos I, Yeung JMC, Arslan J, Carter VM, Isenring E, Kiss N, On Behalf Of The Nourish Point Prevalence Study Group. Assessment of Nutritional Status and Nutrition Impact Symptoms in Patients Undergoing Resection for Upper Gastrointestinal Cancer: Results from the Multi-Centre NOURISH Point Prevalence Study. Nutrients. 2021 Sep 24;13(10):3349. doi: 10.3390/nu13103349. PMID 34684353